CLINICAL TRIAL: NCT02622672
Title: Water-soluble Ubiquinol (a Reduced Form of Coenzyme Q10) Supplementation on Blood Glucose, Lipids, Oxidative Stress, and Inflammation in Patients With Type 2 Diabetes
Brief Title: Water-soluble Ubiquinol Supplementation on Blood Glucose, Lipids, Oxidative Stress, and Inflammation in Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yeh (Other)
Responsible Party: Sponsor-Investigator, Yeh, Principal Investigator, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CS2-15095
Record Dates: First submitted 2015-11-19; First posted 2015-12-04 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Diabetes
Keywords: Antioxidation; Anti-inflammation; Blood glucose; Blood lipids
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Experimental): glycerin.soy-lecithin, and water
  Interventions: Dietary Supplement: Placebo
- Supplement (Experimental): water-soluble Ubiquinol 100 mg/d
  Interventions: Dietary Supplement: water-soluble ubiquinol

INTERVENTIONS:
Dietary Supplement: water-soluble ubiquinol — 100 mg/d
  Other Names: water-soluble coenzyme Q10
  Arms: Supplement
Dietary Supplement: Placebo — glycerin.soy-lecithin, and water
  Arms: Placebo

SUMMARY:
Diabetes is considered an oxidative stress and a chronic inflammatory disease. Coenzyme Q10 (ubiquinone) is recognized as a lipid soluble antioxidant. Ubiquinol is a reduced form of coenzyme Q10 in our body after food or supplements intakes. Studies have indicated that the water-soluble ubiquinol had better antioxidant activity and absorption than lipid-soluble. The purpose of this study was to investigate the effects of a water-soluble ubiquinol supplement (100 mg/d) on antioxidation and anti-inflammation in diabetes patients.

DETAILED DESCRIPTION:
The patients with type 2 diabetes will recruit as subjects (n = 50) and randomly assign to the placebo (n = 25) or coenzyme Q10 groups (n = 25). The intervention will administer for 12 weeks. The concentrations of coenzyme Q10, oxidative stress marker (malondialdehyde), antioxidant enzymes activities (superoxide dismutase, catalase, and glutathione peroxidase), inflammatory markers [C-reactive protein (CRP), and interleukin-6 (IL-6)], and biochemical parameters (fasting glucose, A1C, insulin, C-peptide, and lipid profiles), and blood pressure will measure. Hopefully, the results of this study could provide the information of water-soluble ubiquinol supplement for clinical doctors and dietitians recommend that diabetes patients deserve to know whether the use of coenzyme Q10 supplement.

ELIGIBILITY:
Inclusion Criteria:

* The diagnostic criteria for type 2 diabetes were defined as a glycohemoglobin (A1C) ≧ 6.5%, a fasting glucose ≧ 7.0 mmol/L or a 2-h plasma glucose ≧ 200 mmol/L during an oral glucose tolerance test (OGTT), as well as the use of anti-hyperglycemic drugs.

Exclusion Criteria:

* pregnant or lactation women.
* patients with liver or renal disease
* Antioxidant dietary supplements user.
* patients under warfarin therapy.
* patients with hypoglycemia (fasting glucose < 60 mg/dL) or hyperlipidemia (fasting triglyceride ≧ 500 mg/dL)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | 12 weeks
  serum level of fasting glucose in mmol/L.

SECONDARY OUTCOMES:
Low density lipoprotein-cholesterol (LDL-C) | 12 weeks
  serum level of LDL-C in mmol/L.
high density lipoprotein-cholesterol (HDL-C) | 12 weeks
  serum level of HDL-C in mmol/L.
malondialdehyde (MDA) | 12 weeks
  plasma level of MDA in micromol/L.
catalase (CAT) | 12 weeks
  red blood cells level of CAT in Units/mg protein.
superoxide dismutase (SOD) | 12 weeks
  red blood cells level of SOD in Units/mg protein.
glutathione peroxidase (GPx) | 12 weeks
  red blood cells level of GPx in Units/mg protein.
high sensitivity C-reactive protein (hs-CRP) | 12 weeks
  serum level of hs-CRP in mg/L.
high sensitivity interleukin (hs-IL-6) | 12 weeks
  serum level of hs-IL-6 in pg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Ting Lin, Ph.D., Principal Investigator — School of Nutrition, Chung Shan Medical University